CLINICAL TRIAL: NCT00579319
Title: Use of Breast MRI for Local Staging
Status: Withdrawn | Type: Observational
Why Stopped: There were no subjects ever enrolled. Study was closed at the IRB.
Sponsor: University of Arkansas (Other)
Responsible Party: Steven E. Harms, MD, UAMS
Other Study IDs: 37639
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
When breast MRI is used to determine the extent of local disease, the management changes, resulting in improved outcomes. Studies have indicated that breast MRI plus mammography is better for detecting tumors. surgeons are now utilizing breast MRI to determine the extent of disease in women diagnosed with breast cancer. It has not been established how management of breast cancer patients has been affected by the use of breast MRI or how that management has affected the outcome for these patients. This retrospective chart review will document management and outcome for breast cancer patients who have had pre treatment breast MRI.

DETAILED DESCRIPTION:
When breast MRI is used to determine the extent of local disease, the management changes, resulting in improved outcomes. Studies have indicated that breast MRI plus mammography is better for detecting tumors. surgeons are now utilizing breast MRI to determine the extent of disease in women diagnosed with breast cancer. It has not been established how management of breast cancer patients has been affected by the use of breast MRI or how that management has affected the outcome for these patients. This retrospective chart review will document management and outcome for breast cancer patients who have had pre treatment breast MRI.

The medical records of patients who received breast MRI for pre-treatment staging of breast cancer will be retrospectively reviewed to see if the MRI information affected management. UAMS surgeons will be asked if the breast MRI resulted in:

1. no change in management
2. Moderate change in management-what (modified lumpectomy-larger or smaller)
3. Significant change-what (contralateral breast, additional quadrants, lump to mast, neoadjuvant chemo)-note less dz than w/o MRI, more dz than w/o MRI. The medical record of patients who were imaged will be reviewed for presenting symptom, clinical exam, imaging studies (mammogram, breast ultrasound, breast MRi) and pathology results. This study is limited to retrospective chart review with the only foreseeable risk being that of disclosure of PHI. To minimize this risk, data collection forms will be identified by subject ID number. A master list of these ID numbers linked to subject medical record number will be maintained in the investigator's file and kept in a secure location accessible only to the study team for purposes of verification of data and validation of results. The medical record number will not be recorded on any other form containing subject PHI. The only foreseeable breach of confidentiality would be for the security of the investigator's files to be compromised.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone a breast MRI for staging

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing breast MRI at a community practice in Northwest Arkansas
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-04; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Breast MRI will have a significant impact on patient management | at time of staging

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Harms, MD, Principal Investigator — UAMS